CLINICAL TRIAL: NCT05466227
Title: Improving the Care Trajectory for Patients With Paroxysmal Supraventricular Tachycardia in the Emergency Department by Implementing the Modified Valsalva Maneuver: A Realist Evaluation
Brief Title: Modified Valsalva Maneuver: A Realist Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Pieter Jan Van Asbroeck, MD, Ziekenhuis Oost-Limburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Z-2022052
Record Dates: First submitted 2022-07-05; First posted 2022-07-20 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Supraventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Supraventricular

STUDY DESIGN:
Intervention Model Description: This is a mixed-methods study that uses realist evaluation as the overall conceptual framework to examine a quality improvement program to improve the care for patients with paroxysmal supraventricular tachycardia in the emergency department.
  A realist evaluation is methods-neutral, and the use of a mixed-methods approach employing a case note review, interviews, and focus groups with patients and staff will generate and analyse both qualitative and quantitative data to achieve the goal of the evaluation. Analysis of qualitative and quantitative data will be carried out using a convergent mixed-methods approach to ensure continuous triangulation of multiple data, which will provide a greater understanding of the findings in relation to policy and practice. Broadly, the evaluation could also be considered a process and outcome evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementing Modified Valsalva (Experimental): Implementing Modified Valsalva
  Interventions: Other: Implementation of Modified Valsalva maneuvre

INTERVENTIONS:
Other: Implementation of Modified Valsalva maneuvre — Modified Valsalva maneuvre:
  * Patient is attached to 12-lead ECG monitoring
  * The patient sits in an upright position and performs forced expiration for 15 seconds by blowing on a 10 mL syringe
  * Patient's legs are elevated (45°) for 15 seconds
  * Afterwards, the patient is placed back in an upright position
  * If not efficient, this maneuver can be repeated up to two times

SUMMARY:
Cardiac arrhythmia, specifically paroxysmal supraventricular tachycardia (SVT), accounts for a substantial proportion of emergency medical services resources utilization. Restoring a normal sinus rhythm (reconversion) should be done quickly and effectively. Reconversion requires increasing the atrioventricular node's refractoriness, which can be achieved by vagal maneuvers, pharmacological agents, or electrical cardioversion.

The Valsalva Maneuver (VM) is a commonly used non-invasive reconversion method. It increases myocardial refractoriness by increasing intrathoracic pressure for a brief period, thus stimulating baroreceptor activity in the aortic arch and carotid bodies, resulting in increased parasympathetic (vagus nerve) tone. The effectiveness of conventional vagal maneuvers in terminating SVT, when correctly performed, shows a considerable variation ranging from 19.4% to 54.3%. To improve the effectiveness of the Valsalva Maneuver, the Modified Valsalva Maneuver (MVM) was introduced. While the standard VM is performed when the patient is in a sitting position (45°-90°), the modified VM involves having the patient sit up straight and perform a forced expiration for about 15 seconds, after which the patient is brought into a supine position with the legs raised (45°) for another 15 seconds. This modification should increase relaxation, phase venous return, and vagal stimulation. A recent meta-analysis demonstrated a significantly higher success rate for reconversion to sinus rhythm when using the MVM compared to the standard VM in patients with an SVT (Odds Ratio = 4.36; 95 percent c.i. 3.30 to 5.76; P < .001). More adverse events were reported in the MVM group, although this difference is not significant (Risk Ratio = 1.48; 95 percent c.i. 0.91 to 2.42; P = .11). The available evidence suggests that medication use was lower in the MVM group than in the standard VM group. However, medication use could not be generalized across the different studies. None of the included studies in this review showed a significant difference in length of stay in the emergency department (ED). Hence, the gain of implementing MVM is a higher rate of success with non-invasive reconversion methods. While the available evidence is highly suggestive of supporting the use of the MVM compared to the standard VM in the treatment of adult patients with SVT, implementation seems difficult.

Current evaluations, such as the 'gold-standard' randomised controlled trial (RCT) design, rarely adequately or even explicitly address the context-specific drivers behind implementation outcomes and their relationship to the underlying programme theory, making it difficult to interpret their findings in light of other programmes in different settings. As a result, few evaluation strategies are widely accepted as appropriate. The net benefit of interventions and understanding how variable outcomes are achieved remains empirically uncertain. Therefore, it is essential to develop comprehensive, rigorous, and practical methods to evaluate people-centred quality improvement programmes, inform the selection of effective and efficient interventions, and facilitate improvement and scaling-up. In evaluating such complex interventions, the Medical Research Council (MRC) argues for the importance of process evaluation in conjunction with outcome evaluation to account for variability in implementation. The MRC's process evaluation framework guides evaluators to understand the implementation processes (what is implemented and how), mechanisms of intervention (how the delivery of the intervention produces change) and contextual factors that affect implementation and outcomes.

Research question This study aimed to evaluate a quality improvement program to improve the non-invasive care for patients with paroxysmal supraventricular tachycardia in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients that present to the emergency department
* Only true SVT will be included.

Exclusion Criteria:

* ECG more suggestive of atrial fibrillation or atrial flutter
* Age < 18 years or > 70 years
* Broad QRS, including known aberration
* Known aneurysm (aortic, intracranial or elsewhere)
* Known aortic stenosis
* Known glaucoma
* Hemodynamic instability requiring immediate electric cardioversion.
* Patients that experience an SVT in the hospital but are never admitted to the emergency department (e.g., patients in the cardiac care unit), as the MVM protocol will be only implemented in the prehospital setting and ED.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Was Modified Valsalva maneuver used in this patient? | Moment of treatment, no follow up. Up to 1 year since start of the study.
  Yes/No. Was the patient's supraventricular tachycardie treated with Modified Valsalva or did they use a different treatment?

SECONDARY OUTCOMES:
Was there a need for the use of medication or was the Modified Valsalva maneuver sufficient? | Moment of treatment, no follow up. Up to 1 year since start of the study.
Length of stay in the ED | Moment of treatment, no follow up. Up to 1 year since start of the study.
  How long did the patient stayed in the emergency department?
Adverse events | Moment of treatment, no follow up. Up to 1 year since start of the study.
  Where there any adverse events correlated to the treatment used?
Hospital admission | Moment of treatment, no follow up. Up to 1 year since start of the study.
  Was there a need to admit the patient to the hospital?
Patient experience | Moment of treatment, no follow up. Up to 1 year since start of the study.
  Is it the first time you experienced this rhythm disturbance? To your knowledge, did they treat you by medication, or did they have you do a special maneuver?
  If they have made you do a special maneuver:
  * Can you describe what maneuver they made you do?
  * How many times did you do this maneuver?
  * Was it successful?
  * How did you experience this treatment?
  If they used medication for your rhythm disturbance:
  * How many times did they give you this medication?
  * How did you experience this treatment? If you were treated both by a maneuver and the medication, how did you experience one versus the other?
Staff experience | Moment of treatment, no follow up. Up to 1 year since start of the study.
  Do you know the recently implemented protocol of modified Valsalva maneuver in the treatment of an SVT? Did you use a non-pharmacological maneuver for termination of the SVT?
  * Yes/No
  * If you did not use a non-pharmacological maneuver, explain why.
  * If you did use a non-pharmacological maneuver:
    * What maneuver did you use?
    * Can you describe it step by step? How many times did you apply this maneuver before it was successful or before you stopped trying it?
  * Was it successful?
  * If it was not successful, what was your next step? Did you use medication for the SVT?
  * Yes/No
  * What medication did you use?
  * How many times did you have to give this medication?
  * Was it successful? According to your experience, how do you rate the crowding of the ED on a Likert scale of 0-10?
Efficiency | Moment of treatment, no follow up. Up to 1 year since start of the study.
  Was the supraventricular tachycardia terminated after the used treatment (modified valsalva, valsalva, medication)?

CONTACTS AND LOCATIONS:
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: Undecided